CLINICAL TRIAL: NCT06072820
Title: Analytical Evaluation of the Endotest® Diagnostic
Acronym: ENDORepro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ZIWIG (Industry)
Collaborators: Monitoring Force Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-03
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Endometriosis; Diagnosis
Keywords: Endometriosis; Diagnosis; Saliva sample; Repeatibility; Circadian cycle; Interferences; Stability
MeSH Terms: conditions — Endometriosis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Research Planning (Other): Study population will be composed of subject with a confirmed or ruled-out diagnosis of endometriosis. The subject diagnosis could be ascertained through imaging and/or surgery with or without biopsies.
  After a first assessment during a routing care visit, the subject will be asked to come back for a day, or half a day depending on the impact of the circadian cycle.
  Interventions: Device: Salivary Sampling

INTERVENTIONS:
Device: Salivary Sampling — Inclusion visit: After signature of the informed consent, all subjects will perform 3 consecutive Endotest® Diagnostic during the visit and 1 at-home.
  Circadian circle visit: 6 included subjects will be asked to come back for a full day. They will have to perform 17 Endotest® Diagnostic: 14 on study site and 3 at home after the visit.
  Repeatability-intermediate fidelity-stability-interferences visit: a maximum of 16 included subjects will be asked to come back for this visit. They will have to perform 17 Endotest® Diagnostic: 14 on study site and 3 at home after the visit.

SUMMARY:
This is an interventional with minimal risks and constraints (RIPH 2 in France), prospective, longitudinal, non-randomized, multicenter study.

The present study will allow us to evaluate multiple factors assessing the Endotest® Diagnostic accuracy and its possible limitations. To characterize the Endotest® Diagnostic, the following parameters will be evaluated:

* Repeatability: the verification of the invariability of its results without condition changes,
* Circadian cycle: whether the circadian cycle affects the determination of the signature,
* Intermediate fidelity: the verification of the invariability of its results with an operator change,
* Interferences: the impact of different interferences on its results,
* Stability: the possible modification of its results depending on the samples conditions of storage.

The acts and procedures performed in this research will be divided into three visits:

* Inclusion visit: performance of 4 Endotest® Diagnostics (3 at the visit and 1 at home) by the 60 included subjects,
* "Circadian cycle" visit: performance of 17 Endotest® Diagnostics (14 at the visit and 3 post-visit at home) by 6 subjects selected after evaluation of the results of the inclusion visit,
* "Repeatability-intermediate fidelity-interference-stability" visit: realization of 17 Endotest® Diagnostic by 10 or 16 subjects, depending on the results of the impact of the circadian cycle on the saliva signature. These subjects will be selected according to the results of the inclusion visit, excluding those who participated in the circadian cycle visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 years to 43 years,
* Subject having dated and signed the consent form,
* Subject affiliated to the French health system,
* Subject able to return for a full day for the rest of the study,
* Subject whose diagnosis of endometriosis has been established with certainty or definitively ruled out.

Non-Inclusion criteria:

* Pregnant subject,
* Subject with an acute or chronic infection (viral hepatitis, HIV...),
* Subject with history of hypersensitivity or allergy,
* Subject with a personal history of cancer,
* Subjects with significant difficulties in reading or writing the French language,
* Subject unable to comply with the study and/or follow-up procedures,
* Subject who has objected to the collection of her data,
* Subject participating in an interventional study or in the exclusion period of an interventional study.

Exclusion Criteria:

* Pregnant subject,
* Subject with acute or chronic infection (viral hepatitis, HIV...),
* Subject unable to comply with study and/or follow-up procedures (including absence of outside salivary sample after the inclusion visit),
* Subject participating in an interventional study or in the exclusion period of an interventional study.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Analytical assessment of the Endotest® Diagnostic and result of the Endotest® Diagnostic: positive, negative, inconclusive, not assessable | Through the end of repeatibility study, an average of 3 months
  To evaluate the repeatability of Endotest® Diagnostic (analytical method and signature)
Change from baseline in the result (Yes/No) of the Endotest® Diagnostic | Through the end of repeatibility study, an average of 3 months
  o evaluate the repeatability of Endotest® Diagnostic (analytical method and signature)

SECONDARY OUTCOMES:
Analytical assessment of the Endotest® Diagnostic and result of the Endotest® Diagnostic: positive, negative, inconclusive, not assessable | Through the end of repeatibility study, an average of 3 months
  To evaluate the absence of variation during the day of the results of the Endotest® Diagnostic
Change from baseline in the result (positive/negative) of the Endotest® Diagnostic | Through the end of repeatibility study, an average of 3 months
  To evaluate the absence of variation during the day of the results of the Endotest® Diagnostic
Analytical assessment of the Endotest® Diagnostic and result of the Endotest® Diagnostic: positive, negative, inconclusive, not assessable | Through the end of repeatibility study, an average of 3 months
  To evaluate the intermediate fidelity of the Endotest® Diagnostic (analytical method and signature)
Change from baseline in the result (positive/negative) of the Endotest® Diagnostic | Through the end of repeatibility study, an average of 3 months
  To evaluate the intermediate fidelity of the Endotest® Diagnostic (analytical method and signature)
Analytical assessment of the Endotest® Diagnostic and result of the Endotest® Diagnostic: positive, negative, inconclusive, not assessable | Through the end of repeatibility study, an average of 3 months
  To evaluate the stability of the samples once they are collected
Change from baseline in the result (positive/negative) of the Endotest® Diagnostic | Through the end of repeatibility study, an average of 3 months
  To evaluate the stability of the samples once they are collected
Analytical assessment of the Endotest® Diagnostic and result of the Endotest® Diagnostic: positive, negative, inconclusive, not assessable | Through the end of repeatibility study, an average of 3 months
  To evaluate the absence of interference on the analytical method and the signature
Change from baseline in the result (positive/negative) of the Endotest® Diagnostic | Through the end of repeatibility study, an average of 3 months
  To evaluate the absence of interference on the analytical method and the signature

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Tivoli, Bordeaux, Gironde
  - CHU de Rouen, Rouen, Seine-Maritime